CLINICAL TRIAL: NCT04829253
Title: Effectiveness of a Short and Telematic Version of Cognitive-behavioral Treatment for Borderline Personality Disorder: an Open-label, Non-inferiority Randomized Clinical
Brief Title: Effectiveness of a Short and Telematic Version of Cognitive-behavioral Treatment for Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: University Diego Portales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 210330008
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not be therapists in the study and will be blind to treatment allocation. The only exception involves assessors in charge of evaluating care usage (e.g. ER visits and inpatient) as they will probably find out the treatment condition. These assessors will not participate in the assessment of primary or other secondary outcome measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- b-DBT (Brief Dialectical Behavioral Therapy) (Experimental): 3 months of and intensive modified DBT intervention.
  Interventions: Behavioral: Dialectical Behavior Therapy -3-months
- s-DBT (standard Brief Dialectical Behavioral Therapy) (Active Comparator): 6 months of a standard DBT intervention (this is a shorter version of the original 12-month DBT, but includes all four active components delivered over 6 months)
  Interventions: Behavioral: Dialectical Behavior Therapy -6-months

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy -3-months — Modification of affect regulation, behavioral regulation, interpersonal functioning and identity functioning through the use of skills training, phone check-ins, crisis management and individual initial assessment.
  Arms: b-DBT (Brief Dialectical Behavioral Therapy)
Behavioral: Dialectical Behavior Therapy -6-months — Modification of affect regulation, behavioral regulation, interpersonal functioning and identity functioning through the use of skills training, individual psychotherapy, coaching calls and treatment-team consultation.
  Arms: s-DBT (standard Brief Dialectical Behavioral Therapy)

SUMMARY:
Standard Dialectical Behavioral Therapy (DBT)is an effective treatment for Borderline Personality Disorder (BPD), particularly for patients with significant behavioral and affective dysregulation, including suicidality. However, DBT in its original format is delivered in 12 months, and even though currently there are shorter versions of the treatment being developed and tested, in the context of public mental health care in Chile a shorter, intensive and lighter version of the treatment is likely needed to help patients seeking help for BPD symptoms. This study will test whether a 3 month, intensive and simplified version of DBT is at least equivalent to standard six months DBT with all its components (skills training, individual therapy, coaching calls, and treatment-team consulting). 120 patients diagnosed with BPD we'll be randomly assigned to receive either the short, intensive 3-month intervention or the longer standard 6-month DBT intervention. Baseline measures will be taken pre-treatment, upon treatment completion, and at a 4-month follow-up. Session-to-session change in BPD symptoms will also be measured throughout the treatments. Primary outcomes for the study are BPD symptoms, frequency, and intensity of suicidal activity. Secondary outcome measures include depression scores, quality of life, and ER visits, and days in inpatient care.

ELIGIBILITY:
Inclusion Criteria:

* BPD diagnosis according to DSM-IV criteria, evaluated through a SCID-II structured interview.
* History of suicide attempt or self-harm operationalized as at least two episodes of suicide or self-harm in the last 24 months
* Provide signed informed consent to participate in the study.
* Participant has not received more than 8 weeks of DBT in the past 24 months.

Exclusion Criteria:

* Fulfill diagnostic criteria for psychotic disorders classified in ICD-10 (F20-F29), evaluated through the MINI interview.
* Diagnosis of Antisocial Personality Disorder evaluated through the SCID-II.
* Active substance use disorder within the last 3 months, assessed by ASSIST.
* Harmful use or problem dependence on alcohol assessed through AUDIT.
* Meet criteria for Bipolar Affective Disorder type I assessed through the MINI Mania module.
* Significant cognitive impairment assessed through Moca (Moca> 21).
* Diagnosis recorded in the clinical record of intellectual-cognitive disability.
* Recording in the clinical record of medical or surgical problems that could imply a probable hospitalization within one year of the start of the study (for example, cancer, coronary heart disease, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Change in Borderline Personality Disorder Symptoms as measured by the Zanarini Rating Scale for Borderline Personality Disorder - ZAN-BPD | Administered pre-treatment and then weekly until 3 months or 6 months depending on thr study arm. Follow-up assessment at month 7 or month 10 depending on study arm.
  We will capture incremental change in affect dysregulation, behavioral dysregulation, interpersonal functioning, and cognitive/self functioning
Change in the intensity and frequency of suicidal and self-harming activity, measured by a Spanish version of the Suicide Attempt Self-Injury Interview (SASII) | Administered pre-treatment and then at treatment completion, which is at the 3 month mark or 6 month mark depending on thr study arm. Follow-up assessment at month 7 or month 10 depending on study arm.
  Assessment recovers detailed information about frequency, topography, severity, social context, intent, precipitating events, concurrent events and outcomes of suicidal and self-harming behavior during a three-month period.

SECONDARY OUTCOMES:
Depression Symptomatology measured through the Patient Health Questionnaire - PHQ-9 | Administered pre-treatment and then at treatment completion, which is at the 3 month mark or 6 month mark depending on thr study arm. Follow-up assessment at month 7 or month 10 depending on study arm.
  Self-assessment of DMS-IV symptoms of depression.
Reasons for Living measured though the RFL | Administered pre-treatment and then at treatment completion, which is at the 3 month mark or 6 month mark depending on thr study arm. Follow-up assessment at month 7 or month 10 depending on study arm.
  Self-report scale that measures reasons an individual has to live and thus prevents him/her from potentially engaging in suicidal activity
Quality of life measured through the World Health Organization Quality of Life brief version; WHOQOL-BREF | Administered pre-treatment and then at treatment completion, which is at the 3 month mark or 6 month mark depending on thr study arm. Follow-up assessment at month 7 or month 10 depending on study arm.
  Measures overall satisfaction with life
Emergency Room Visit measured by the integrated electronic records. | Administered pre-treatment and then at treatment completion, which is at the 3 month mark or 6 month mark depending on thr study arm. Follow-up assessment at month 7 or month 10 depending on study arm.
  Indicates number of visits to the ER in a target 3 month period as documented in electronic records
Psychiatric inpatient days measured by the integrated electronic records. | Administered pre-treatment and then at treatment completion, which is at the 3 month mark or 6 month mark depending on thr study arm. Follow-up assessment at month 7 or month 10 depending on study arm.
  Indicates number of days spent in psychiatric inpatient care in a target 3 month period as documented in electronic records

CONTACTS AND LOCATIONS:
Overall Officials: Alex Behn, PhD, Principal Investigator — Millennium Institute for Research in Depression and Personality
Locations (1):
- Complejo Asistencial Dr. Sótero del Río, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD at this point.